CLINICAL TRIAL: NCT04420923
Title: A Randomised Controlled Trial Testing the Efficacy of the Treatment Strategy Observe-and-Plan Against Standard Treat-and-Extend in a Population of Newly Referred Patients With Age-related Macular Degeneration.
Brief Title: Optimizing the Treatment Strategy for Age-related Macular Degeneration
Acronym: OnP2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); Molde Hospital (Other); Alesund Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 90953
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Wet Macular Degeneration
Keywords: Outcome Assessment, Health Care
MeSH Terms: conditions — Wet Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observe-and-Plan (Experimental): Patients will follow the same protocol as described by dr. Mantel et al. (2014) in the first Observe-and-Plan study conducted in Lausanne.
  Interventions: Other: Observe and Plan
- Treat-and-Extend (Active Comparator): Patients will follow the standard treatment protocol for Treat-and-Extend, used for several years in the participating clinics.
  Interventions: Other: Treat-and-Extend

INTERVENTIONS:
Other: Observe and Plan — First the individual interval between the injections of anti-VEGF (vascular endothelial growth factor) is established by observing the time from the loading dose to recurrence of the disease. The patient will come to control every four weeks to establish this interval. Second, the patient will receive injections at intervals that are two weeks shorter than the observed period. 2-3 injections are given before the next control. The control should be no later than six months ahead.
  Arms: Observe-and-Plan
Other: Treat-and-Extend — At the first control 4 weeks after the loading dose, the ophthalmologist assesses whether the macula is still wet or whether the macula is dry. In case of wet macula, the patient receives a new injection on the same day and a new control in 4 weeks. If the macula is dry, the patient will return in 2 weeks for the next injection, ie the injection interval is extended from 4 to 6 weeks.
  Patients will be controlled every time they are to receive an intravitreal injection. If the macula is dry, the injection interval will be extended by 2 weeks and if the macula is wet the interval is shortened by 2 weeks. The shortest interval will be 4 weeks.
  Other Names: Standard treatment
  Arms: Treat-and-Extend

SUMMARY:
The purpose of this study is to compare two different treatment protocols for wet macular degeneration; the new protocol called "Observe and Plan" against the current standard protocol "Treat and Extend". Studies suggest that patients achieve equally good visual acuity with fewer controls and that they are more satisfied with the new protocol.

DETAILED DESCRIPTION:
The purpose of the study is to test a new treatment protocol for wet macular degeneration, called "Observe and Plan", against today's standard protocol "Treat and Extend". Studies suggest that the individual treatment interval can be achieved earlier with "Observe-and-Plan" and that a proportion of patients do not need more than 3 injections, ie the loading dose. The other advantages seem to be that patients achieve good visual acuity with fewer controls and are more satisfied with the new protocol, which will be beneficial to both patients and health care. To our knowledge, no randomized controlled trial has tested this before.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed age-related macular degeneration according to criteria.
* new diagnose of active CNV verified with OCTA or FA / ICGA.
* BCVA ≥ 20/200 measured with ETDRS visual acuity chart
* written informed consent

Exclusion Criteria:

* Eyes formerly treated with anti-VEGF, photodynamic therapy, radiation therapy, transpupillary thermotherapy or focal laser photocoagulation involving the macular area.
* Geographic atrophy and subretinal fibrosis affecting the patient's visual acuity.
* Any other ongoing eye disease that influences patient's visual acuity, such as glaucoma with central vision loss, proliferative diabetic retinopathy, diabetic macular edema or chronic uveitis.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2020-05-20 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | 1 year
  Number of letters read at the ETDRS chart will be tested for each eye starting with a test distance of 2 meter, after correction of the refraction. A standardized testing protocol will be used both for refraction and the visual acuity test.
Visual acuity | 2 years
  Number of letters read at the ETDRS chart will be tested for each eye starting with a test distance of 2 meter, after correction of the refraction. A standardized testing protocol will be used both for refraction and the visual acuity test

SECONDARY OUTCOMES:
Patient satisfaction assessed by NEI-VFQ-25 | 1 year
  National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25). The VFQ-25 is a reliable and valid 25-item version of the 51-item National Eye Institute Visual Function Questionnaire (NEI-VFQ). It is especially useful in settings such as clinical trials, where interview length is a critical consideration.
Patient satisfaction assessed by NEI-VFQ-25 | 2 years
  National Eye Institute Visual Function Questionnaire-25 (NEI-VFQ-25). The VFQ-25 is a reliable and valid 25-item version of the 51-item National Eye Institute Visual Function Questionnaire (NEI-VFQ). It is especially useful in settings such as clinical trials, where interview length is a critical consideration.
Number of injections | 1 year
  The number of injections will be counted for each participant.
Number of controls | 1 year
  The number of controls by the ophthalmologist will be counted for each participant.
Number of injections | 2 years
  The number of injections will be counted for each participant.
Number of controls | 2 years
  The number of controls by the ophthalmologist will be counted for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Dordi Austeng, MD PhD, Principal Investigator — Norwegian University of Science and Technology, Fac MH, INB; Marit Fagerli, MD, Study Director — Clinic of Ear-Nose-Throat, Eye and Maxillofacial Surgery, St. Olavs Hospital; Jorunn Helbostad, Professor, Study Director — Norwegian University of Science and Technology, Fac MH, INB
Locations (3):
- Norway (3):
  - Ålesund Hospital, Ålesund
  - Molde Hospital, Molde
  - Dept. of Ophthalmology, St Olavs Hospital, Trondheim University Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD that underlie results in a publication and related data dictionaries available to other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available on request after publication.
Access Criteria: The requests will be evaluated by the research group at the institute.

REFERENCES:
- [Background] Mantel I, Niderprim SA, Gianniou C, Deli A, Ambresin A. Reducing the clinical burden of ranibizumab treatment for neovascular age-related macular degeneration using an individually planned regimen. Br J Ophthalmol. 2014 Sep;98(9):1192-6. doi: 10.1136/bjophthalmol-2013-304556. Epub 2014 Apr 10. PMID 24729031